CLINICAL TRIAL: NCT06753656
Title: Prospective Randomised Controlled Trial Evaluating the Outcomes of Open Reduction-Internal Fixation With Minimally Invasive Percutaneous Plate Osteosynthesis in Lateral Malleolus Fractures
Brief Title: Comparison of Patients Who Underwent Open and Minimally Invasive Fixation in Lateral Malleolar Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Emre Kurt, Principal Investigator, Medical Doctor, Orthopaedics and Traumatology,, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ordu University CREC 2022/229
Record Dates: First submitted 2024-12-18; First posted 2024-12-31 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Lateral Malleolus Fracture; Minimally Invasive Surgical Procedure; Postoperative Pain; Patient Discharge
Keywords: Lateral Malleolus Fractures; Minimally Invasive Surgery; Postoperative Pain
MeSH Terms: conditions — Ankle Fractures; Pain, Postoperative | interventions — Conversion to Open Surgery; Minimally Invasive Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Randomisation was performed before the first patient was included in the study. Patients were numbered according to the order of hospitalisation. According to these numbers, the surgical technique was applied to the patients according to the surgical technique group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be informed about both surgical techniques. Informed consent will be obtained. Accepting patients will be included in the study. Which group the patients are in will be masked. The surgical group in the follow-up will be explained.
  Outcome assessors were masked. Outcome assessors are senior surgeon and radiology doctor. Scoring will be taken by the senior surgeon. Radiological measurements will be performed at different times by the radiology doctor and the senior surgeon.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally Invasive Surgery (Experimental): Closed reduction of the fracture without opening the fracture site
  Interventions: Procedure: Minimally Invasive Surgery
- Open Surgery (Active Comparator): open reduction of the fracture by opening the fracture site
  Interventions: Procedure: Open Surgery

INTERVENTIONS:
Procedure: Open Surgery — Open surgery technique: A longitudinal incision is made over the lateral malleolus, followed by sharp dissection down to the bone. The fracture is reduced under direct visualization and fixed with a plate and screws.
  Arms: Open Surgery
Procedure: Minimally Invasive Surgery — Closed surgery technique: A 2-3 cm longitudinal incision is made distal to the lateral malleolus to allow for plate placement. A periosteal elevator is used to create a pathway for the plate. The fracture is reduced in a closed manner using reduction clamps, and the plate position is confirmed fluoroscopically. A second longitudinal incision is made proximal to the fracture, and the plate is temporarily fixed with Kirschner wires. The plate is then used as an external guide, with screws placed through mini-incisions. The fracture is fixed with the plate-screw system in a minimally invasive manner.
  Arms: Minimally Invasive Surgery

SUMMARY:
The aim of this study was to compare the postoperative clinical, functional and radiological results of two different surgical methods, minimally invasive percutaneous plate osteosynthesis method and open reduction-internal fixation method, for lateral malleolus fractures in patients presenting with ankle fractures.

DETAILED DESCRIPTION:
The study is a prospective randomized controlled clinical trial planned to be conducted at the Republic of Turkey Ministry of Health, Giresun University Faculty of Medicine, Giresun Training and Research Hospital, Department of Orthopedics and Traumatology.

The study includes patients who will undergo surgery for lateral malleolus fractures. No additional tests will be requested outside of routine clinical, radiological, and laboratory evaluations required during surgery, hospitalization, and outpatient follow-ups.

The routine treatment protocol for patients undergoing surgery for lateral malleolus fractures in clinic is as follows:

* A detailed medical history is obtained, followed by systemic and local examinations.
* Radiological evaluations, including comparative ankle radiographs (Anterior-Posterior, Lateral, and Mortise views) and computed tomography (CT) scans, are performed.
* The affected ankle is placed in a splint. Elevation and cold application are performed. Embolism prophylaxis is administered with enoxaparin.
* Anesthesia preparation is performed. The splint is removed daily for examination, and surgery is performed once skin folds are appropriate.
* Post-surgical and outpatient follow-ups include routine ankle radiographs.
* Prophylactic antibiotics are administered preoperatively.
* Analgesics, including paracetamol, non-steroidal anti-inflammatory drugs (NSAIDs), and opioids, are administered based on the patient's pain level, provided there are no contraindications.
* After surgical site monitoring, antibiotic prophylaxis, and analgesia control, the patient is discharged.
* Postoperative follow-ups are scheduled for the 2nd week, 4th week, 6th week, 3rd month, 6th month, and 1st year.
* For the first two weeks postoperatively, dressings are performed every other day, and sutures are removed during outpatient control.
* Patients walk with bilateral crutches non-weight bearing for the first 6 weeks. If syndesmosis screws are used, they are removed with a day-case hospitalization under local anesthesia at the end of the 6th week.
* Partial weight-bearing begins after the 6th week, and the load is progressively increased weekly. Crutches are discontinued 3 months postoperatively.
* Ankle range-of-motion exercises are planned and initiated by the attending surgeon before discharge.
* During outpatient follow-ups, the ankle is re-examined, and any patient complaints are evaluated and managed with appropriate investigations and treatments.

In patients who consent to participate in the study, the following data will be collected:

* Demographic data: Gender, age, education level, occupation, height, body weight, body mass index (BMI), affected side, lateralization, diagnosis, smoking status, alcohol use, comorbidities, and medications.
* Follow-up data: Fracture etiology, time of fracture occurrence, fracture mechanism, soft tissue classification (Ostern-Tscherne), fracture type based on Weber and Lauge-Hansen classifications, preoperative hospitalization duration, time of surgery, type and duration of anesthesia, surgical technique, surgical duration, syndesmosis fixation, tourniquet use (and duration), fluoroscopy frequency and duration, use of drains (and removal time), postoperative hospitalization duration, use of tranexamic acid for bleeding control, discharge date, medications used during hospitalization and post-discharge, postoperative splint use, and syndesmosis screw removal timing if applicable.

Surgical approach:

Patients undergoing lateral malleolus surgery are operated on in the supine position under anesthesia with the hip elevated. A tourniquet is applied. Following the preparation of the lower extremity with povidone-iodine, the surgical method-open or minimally invasive-is selected based on the surgeon's experience.

* In the open approach: A longitudinal incision is made over the lateral malleolus, followed by sharp dissection down to the bone. The fracture is reduced under direct visualization and fixed with a plate and screws.
* In the minimally invasive method: A 2-3 cm longitudinal incision is made distal to the lateral malleolus to allow for plate placement. A periosteal elevator is used to create a pathway for the plate. The fracture is reduced in a closed manner using reduction clamps, and the plate position is confirmed fluoroscopically. A second longitudinal incision is made proximal to the fracture, and the plate is temporarily fixed with Kirschner wires. The plate is then used as an external guide, with screws placed through mini-incisions. The fracture is fixed with the plate-screw system in a minimally invasive manner.
* Regardless of the fixation method, the surgical site is irrigated with saline, incisions are closed with sutures, dressings are applied, and a short-leg splint is used to facilitate soft tissue healing. The operation is then concluded.

Radiological assessment:

Fracture classification will be performed based on direct radiographs. Additionally, radiographic parameters, including medial clear space, tibiofibular overlapping, tibiofibular clear space, talar tilt, and talocrural angle, will be measured and compared with the unaffected ankle.

Planned clinical scoring scales and evaluation timelines:

* Numeric Pain Rating Scale (NPRS): Preoperatively, and postoperatively 8th hour, 24th hour, 2nd week, 4th week, 6th week, 3rd month, 6th month, and 1st year
* AOFAS (American Orthopaedic Foot and Ankle Society) Ankle Score: Postoperatively 3rd month, 6th month, and 1st year

ELIGIBILITY:
Inclusion criteria;

* being a volunteer,
* closed distal fibular epiphysis,
* Lateral malleolus fractures operated for Weber type B or C fractures,
* patients with regular follow-up in outpatient clinic

Exclusion criteria;

* open fractures
* fractures accompanied by pylon fractures,
* fractures accompanied by talus fractures,
* patients with a previous fracture/surgery of the same or another ankle,
* ankles accompanied by arthrosis,
* pathological fractures
* multitrauma or polytrauma patients,
* those with psychiatric or neurological diseases,
* illiterate patients,
* congenital or acquired deformity of the lower extremities
* Patients who could not be reduced intraoperatively closed and who underwent open surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Post operative Pain | Preoperatively and postoperatively 8th hour, 24th hour, 2nd week, 4th week, 3rd month, 6th month and 1st year
  Patients were analysed for pain scores according to the numeric pain rating scale(NPRS) for the following periods
Patient discharge time | Up to 12 months
  Preoperative, postoperative and total hospital stay and discharge times of the patients were recorded.

SECONDARY OUTCOMES:
The number and duration of fluoroscopy | Postoperative 1st day
  The number and duration of fluoroscopies used during the entire surgery for each patient is recorded.
Functional score | Postoperatively 3rd month, 6th month and 1st year
  AOFAS scores were obtained at the follow-up visits of the patients at the following times

CONTACTS AND LOCATIONS:
Overall Officials: Kürşad Aytekin, M.D., Study Director — Giresun University
Locations (1):
- Giresun University Faculty of Medicine-Giresun Training and Research Hospital, Giresun, Turkey (Türkiye)